CLINICAL TRIAL: NCT00002240
Title: Evaluation of the Safety and Antiviral Efficacy of a Novel HIV-1 Protease Inhibitor, BMS-232632, Alone and in Combination With d4T and ddI as Compared to a Reference Combination Regimen
Brief Title: Study of a New Protease Inhibitor, BMS-232632, in Combination With Other Anti-HIV Drugs
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Purpose: Treatment
Other Study IDs: 302A; AI424-007
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2011-05-04 (Estimated); Status verified 2011-04

CONDITIONS: HIV Infections
Keywords: Didanosine; Dose-Response Relationship, Drug; Drug Therapy, Combination; Stavudine; HIV Protease Inhibitors; Reverse Transcriptase Inhibitors; Anti-HIV Agents; Nelfinavir
MeSH Terms: conditions — HIV Infections | interventions — Atazanavir Sulfate; Nelfinavir; Stavudine; Didanosine

INTERVENTIONS:
Drug: Atazanavir
Drug: Nelfinavir mesylate
Drug: Stavudine
Drug: Didanosine

SUMMARY:
The purpose of this study is to evaluate a new protease inhibitor known as BMS-232632. This drug will be given in combination with 2 other anti-HIV drugs (stavudine and didanosine). The effectiveness of BMS-232632 against HIV infection will be compared to that of nelfinavir, a protease inhibitor that is already commonly prescribed.

DETAILED DESCRIPTION:
Patients are randomized to receive one of two drug regimens: BMS-232632, ddI, and d4T or NFV, ddI, and d4T. Three different doses of BMS-232632 are used in this study. Randomization is stratified for HIV RNA level (less than 30,000 copies/ml versus 30,000 or greater copies/ml). Patients remain on their drug regimen for 48 weeks.

ELIGIBILITY:
Inclusion Criteria

Patients may be eligible for this study if they:

* Are HIV-positive.
* Have an HIV blood level between 2,000 and 200,000 copies/ml.
* Have a CD4 cell count of at least 100 cells/mm3.
* Are 18 years of age or older.
* Are available for follow-up for at least 48 weeks.
* Agree to use a barrier method of birth control (such as condoms) during the study.

Exclusion Criteria

Patients will not be eligible for this study if they:

* Have ever received anti-HIV (antiretroviral) treatment.
* Have an HIV-related opportunistic infection or condition at the time of study entry.
* Have primary HIV infection, meaning they have recently been infected.
* Have had severe diarrhea within the 30 days before study entry.
* Have hemophilia.
* Have a history of pancreatitis, hepatitis, or a peripheral neuropathy.
* Are unable to tolerate oral medication.
* Are pregnant or breast-feeding.
* Abuse alcohol or drugs.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 1999-03; Primary Completion 2001-12 (Actual); Study Completion 2001-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (17):
- United States (16):
  - Clinsites / Sorra Research Ctr, Birmingham, Alabama
  - Univ of Alabama at Birmingham, Birmingham, Alabama
  - UCSD Treatment Ctr, San Diego, California
  - UCSF - San Francisco Gen Hosp, San Francisco, California
  - Univ of Colorado / Health Science Ctr, Denver, Colorado
  - ViRx / Dupont Circle Physicians Group, Washington D.C., District of Columbia
  - AIDS Research Consortium of Atlanta, Atlanta, Georgia
  - Rush Presbyterian - Saint Luke's Med Ctr, Chicago, Illinois
  - Washington Univ School of Medicine, St Louis, Missouri
  - Albany Med College, Albany, New York
  - Beth Israel Med Ctr, New York, New York
  - Columbia Presbyterian Med Ctr, New York, New York
  - Case Western Reserve Univ, Cleveland, Ohio
  - Oak Lawn Physicians Group, Dallas, Texas
  - Univ of Texas Southwestern Med Ctr of Dallas, Dallas, Texas
  - Univ TX Galveston Med Branch, Galveston, Texas
- Ottawa General Hospital, Ottawa, Ontario, Canada

REFERENCES:
- [Background] Piliero P, et al. AI424-007: Atazanavir: an HIV protease inhibitor (PI) that does not cause lipid elevations. International Symposium on Drugs Affecting Lipid Metabolism. 2001 Sept 9 - 12
- [Background] Gatell JM, et al. AI424-007: Atazanavir (BMS-232632): Absence of serum lipid changes after 48 weeks of treatment in treatment-naive HIV-positive subjects (Trial AI424007). 8th European Conf on Clinical Aspects and Treatment of HIV Infection (8th ECCATHI). 2001 Oct 28 - 31 (abstract no 223)
- [Background] Piliero P, et al. AI424-007: BMS-232632 - Clinical Trial AI424007: Safety, Efficacy of a Once-Daily Protease Inhibitor at 24 Weeks. 5th International Congress on Drug Therapy in HIV Infection. 2000 Octr 22 - 26
- [Background] Sanne I, Piliero P, Wood R, Kelleher T, Cross A, Mongillo A, Schnittman S. AI424-007: Safety and Antiviral Efficacy of a Novel Once-Daily HIV-1 Protease Inhibitor BMS-232632: Preliminary Results from a Phase II Clinical Trial. 7th Conf Retroviruses and Opportunistic Infect. 2000 Jan 30-Feb 2 (abstract no 672)
- [Background] Squires K, Gatell J, Piliero P, Sanne I, Wood R, Schnittman SM. AI424-007: 48-week safety and efficacy results from a phase II study of a once-daily HIV-1 protease inhibitor (PI), BMS-232632. 8th Conf Retro and Opportun Infect. 2001 Feb 4-8 (abstract no 15)
- [Background] Sanne I, Piliero P, Wood R, Kelleher T, Cross A, Mongillo A, Schnittman S. AI424-007: Safety and Antiviral Efficacy of a Once-Daily HIV-1 Protease Inhibitor BMS-232632: 24 Week Results from a Phase II Clinical Trial. 40th Interscience Conf on Antimicrobial Agents and Chemotherapy. 2000 September 17-20 (abstract no 691)
- [Background] Piliero P, Cahn P, Pantaleo G, Gatell JM, Squires K, Percival L, Sanne I, Wood R, Phanuphak P, Shelton S, Lazzarin A, Thiry A, Kelleher T, Giordano M, Schnittman SM. AI424-007: Atazanavir: A Once-Daily Protease Inhibitor with a Superior Lipid Profile-Results of Clinical Trials Beyond Week 48. 9th Conf on Retroviruses and Opportunistic Infect. 2002 Feb 24 - 28 (abstract no 706-T)